CLINICAL TRIAL: NCT01884025
Title: Get Moving and Get Well: A Behavioral Activation Program for Veterans With SMI
Brief Title: Get Moving and Get Well - Pilot Study
Acronym: GMGWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPO 13-187
Record Dates: First submitted 2013-06-05; First posted 2013-06-21 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression; Post Traumatic Stress Disorder
Keywords: patient centered care; physical activity; behavioral activation; self efficacy; serious mental illness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Motor Activity | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Get Moving and Get Well (Experimental): Walking class developed for Veterans with serious mental illness and administered as part of the PRRC
  Interventions: Behavioral: Get Moving and Get Well
- Health and Humor Class (Sham Comparator): Equally engaging attention control condition
  Interventions: Behavioral: Health and Humor Class

INTERVENTIONS:
Behavioral: Get Moving and Get Well — Walking Class
  Other Names: GMGW
  Arms: Get Moving and Get Well
Behavioral: Health and Humor Class — Class about the role of humor in health
  Other Names: Health and Humor
  Arms: Health and Humor Class

SUMMARY:
Individuals with serious mental illness have greater morbidity from physical illness and mortality than the general population, but tend not to initiate or sustain engagement in health promotion interventions. Although promising weight management and wellness interventions have been developed for this population, they are very intensive and tend to have low enrollment, high attrition, and low reach. This pilot study will investigate a novel low-demand intervention that may be initially more acceptable, the Get Moving and Get Well! (GMGW) program. The primary objectives of the proposed study are to investigate the effects of participation in the GMGW program on measures of behavioral activation, self-efficacy, physical activity, general physical and mental health, mood, participants' intent to engage in more intensive physical health interventions, and actual engagement in those programs. Results of this pilot study will inform a future full-scale study of GMGW.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare: Individuals with serious mental illness (SMI) have greater physical illness morbidity and mortality than the general population, but typically do not enroll in nor complete health promotion interventions. This pilot study will provide preliminary evaluation of a low-demand physical activity intervention that may be acceptable to Veterans with SMI and lead to improved health in this medically vulnerable population.

Project Background: The relatively high rates of morbidity and mortality found among individuals with SMI have led to prioritization by Mental Health QUERI, and other groups, of prevention and health promotion in addition to improved coordination of physical health care for this population. Although promising health promotion interventions have been developed, they are intensive and none seem to successfully address the challenge of improving reach and enrollment while minimizing attrition. We propose to conduct a pilot evaluation of a novel low-demand intervention that may be an acceptable introduction to health promotion, the Get Moving and Get Well! (GMGW) program. Participants in the current version of GMGW have described benefits beyond those expected. We believe a 12-week GMGW program may be an effective and relatively low-demand intervention to promote self-efficacy and physical health in Veterans with SMI through increasing Veteran behavioral activation.

Project Objectives: The objectives of the proposed study are to: (a) determine the effects of participation in the 12-week GMGW program on a measure of behavioral activation; (b) determine the effects of GMGW on measures of self-efficacy, physical activity, general physical and mental health, and mood; and (c) determine the effects of participation in the class on measures of intent to engage and actual engagement in more intensive physical health programs.

Project Methods: In order to inform a future full scale study, we will complete the development of a 12-week manualized GMGW class, assess its acceptability, feasibility and time burden, and evaluate effects of the intervention on key outcome measures. To achieve the aims of the study, we will randomly assign 30 participants to either GMGW or an attention control condition. Participants will complete baseline measures investigating behavioral activation, self-efficacy, physical activity, physical and emotional health, mood, and intent to engage in health promotion activities before beginning the class. These measures will be repeated at the end of the 12-week class, along with questions investigating the acceptability of the interventions. A chart review will investigate actual engagement in health promotion interventions. We will be looking for the emergence of trends for differences in expected directions and response patterns within and between groups that will inform us about effect sizes for the measures and permit a power analysis for the full scale trial. We plan to use repeated measures analysis of variance, controlling for any variables that differ significantly between the intervention and control groups, to test the hypothesis that GMGW participants will have greater improvements on the measures at the end of the 12-week intervention than the control participants. Finally, we will also compare the number of participants who have evidence of participation in new health promotion activities in their medical record using a chi-square test of equal proportions.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for participation, potential participants must be Veterans at the Central Arkansas Veterans Healthcare System.
* They must express an interest in improving their physical health but not be referred to MOVE! at the time of enrollment in the study;

  * not have attended more than six class sessions of GMGW in the past; agree to be randomized to one of two treatment groups (GMGW or control health promotion class);
  * be between the ages of 18 and 65; speak and understand English;
  * and be able to increase walking and light to moderate physical activity as indicated by a progress note by their primary care provider.
* Participants must meet PRRC admission criteria for serious mental illness (primary diagnosis of psychotic disorders,

  * bipolar disorder, major depression and/or severe PTSD) and
  * dysfunction (Global Assessment of Functioning (GAF) score of 50 or less); this will be assessed though a review of the Veteran's CPRS electronic record.

Exclusion Criteria:

* We will exclude Veterans who have been found to be legally incompetent or have a legal guardian of person.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Viverito, PsyD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Get Moving and Get Well | Health and Humor Class
Started | 13 | 14
Completed | 10 | 10
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed both baseline and follow-up measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Get Moving and Get Well | Health and Humor Class | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (6.77) | 54.1 (8.8) | 54.6 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (Non-Hispanic) | 6 | 6 | 12
  African American | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Years of Education [Number; unit: participants]
  HighSchool/GED | 4 | 4 | 8
  Some COllege | 4 | 2 | 6
  Bachelors Degree | 2 | 2 | 4
  Graduate Degree | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Activation for Depression Scale
Description: The BADS asks respondents to rate how much the statements are true for four subscales: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment. It has been found to have acceptable internal consistency (Cronbach's alpha of .87), test-retest reliability (Pearson's r = .74), good construct validity, and when administered to a clinically depressed sample, the factors held up. Items for each subscale are summed to generate subscale scores. The BADS is made up of 25 questions with response option range from 0 (not at all) to 6 (completely). (Subscore Ranges: Activation: 0-108, Avoidance/Rumination: 0-102, Work/School Impairment: 0-120, Social Impairment: 0-120 Total: 0-150). For all subscales, high scores are consistent with the scale name.
Time Frame: Baseline (Time point 0 - Pre intervention/control class) and follow-up (Time point Week 12 - after completion of intervention/attention control class)
Population: Analysis population includes participants who completed both baseline and follow-up measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale
  Activation | 1.3 (6.11) | 1.2 (8.90)
  Avoidance/Rumination | 2.8 (10.25) | 3 (9.76)
  Work/School Impairment | 4.8 (6.27) | 12 (6.05)
  Social Impairment | 3.6 (5.8) | 1.1 (5.51)
  Total Score | 12.5 (21.99) | 6.5 (26.31)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in total BADS score; Test type: Superiority or Other; p = 0.59, t-test, 2 sided; t-Value: 0.55
Statistical Analysis 2: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in Activation Subscale; Test type: Superiority; p = 0.98, t-test, 2 sided; t Value: 0.03
Statistical Analysis 3: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in Avoidance/Rumination Subscale; Test type: Superiority; p = 0.96, t-test, 2 sided; DF: 18 1 Value: -0.04
Statistical Analysis 4: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in Work/School Impairment Subscale; Test type: Superiority; p = 0.21, t-test, 2 sided; t Value: 1.31
Statistical Analysis 5: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in Social Impairment Subscale; Test type: Superiority; p = 0.34, t-test, 2 sided; t Value: 0.99

2. Secondary Outcome: Change in Exercise Self-Efficacy Questionnaire
Description: Based on the exercise self-efficacy factors of resisting relapse and making time for exercise, the Exercise Self-Efficacy questionnaire asks respondents to circle how confident they are about their ability to exercise under difficult conditions, such as "when I am tired". An additional item will be added to include hot weather as a possible barrier to physical activity, because of the likelihood of high spring and summer temperatures in our location. This scale was found to be highly reliable (test-retest reliability was .90) (Markus et al., 1992). It is made up of six questions each on a likert-type scale ranging from 1 (not at all confident) to 7 (very confident). These are ratings are then summed for the total score; total score ranges from 6-42 with higher scores indicating higher exercise self efficacy.
Time Frame: as for outcome 1
Population: Analysis population includes participants who completed both baseline and follow-up measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | 1.5 (4.90) | .6 (6.7)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = 0.75, t-test, 2 sided; t Value: 0.33

3. Secondary Outcome: Change in CHAMPS (Community Healthy Activities Model Program for Seniors) Questionnaire for Older Adults - Physical Activity Frequency
Description: Physical activity and cognitive/social activity will be measured by the CHAMPS (Stewart, et al., 2001) which asks respondents to identify if they participated in an activity (yes or no) how many times a week they participated (continuous variable) and if they did participate, for how many hours per week (rated on a six point scale ranging from less than one hour to more than 9 hours). The CHAMPS assesses for both physical and social/cognitive activities (e.g., "Visit with friends or family (other than those you live with);" "walk briskly").
Time Frame: baseline and 12 week follow-up
Population: Participants who completed baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
times per week
  Physical Activity Frequency | 2.7 (11.84) | 4.3 (7.53)
  Moderate Physical Activity Frequency | 1.3 (5.42) | 2.1 (3.51)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in overall physical activity frequency were compared between the two groups; Test type: Superiority or Other; p = 0.72, t-test, 2 sided; t Value: -0.36
Statistical Analysis 2: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in moderate physical activity frequency between the two groups; Test type: Superiority; p = 0.70, t-test, 2 sided; t Value: -0.39

4. Secondary Outcome: Change in Veterans RAND 12 (VR-12)
Description: The VR-12 is based on the Veterans RAND 36 (SF-36) and has been shown to be a good outcome measure of general physical and mental health with significant correlations with morbidity (Kazis, et al., 2006). It provides physical and mental health subscale scores. It consists of 12 questions (several with sub sections) which are rated on three point and five point likert-type scales. These ratings are then assigned values with some scored opposite so that higher values always indicate more positive health. The Physical Health component can range from 10-59 and the Mental Health component from 6-33.
Time Frame: Baseline and Follow -up
Population: Participants who completed both baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale
  Physical Health | 0.54 (9.033) | -2.5097 (8.74)
  Mental Health | 7.52 (12.75) | 3.31 (11.86)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in the physical health scale of the RAND 12 were compared; Test type: Superiority; p = 0.45, t-test, 2 sided; t Value: 0.77
Statistical Analysis 2: Comparison: Get Moving and Get Well vs Health and Humor Class; Change in the mental health scale of the RAND 12 were compared; Test type: Superiority; p = 0.45, t-test, 2 sided; t Value: 0.76

5. Secondary Outcome: Change in Personal Health Information Depression Scale (PHQ-8)
Description: Depression will be measured by the Patient Health Questionnaire-8 (PHQ-8) which has been validated across several populations (Kroenke & Spitzer, 2002). Respondents rate how often they were bothered by eight problems on a likert-type scale ranging from 0 (not at all) to 3 (nearly every day). Scores can range from 0-24; higher scores indicate higher levels of depression with score >10 indicating clinically relevant depression.
Time Frame: Baseline and Follow-up
Population: participants who completed both baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | -1.30 (5.14) | -.50 (4.72)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority or Other; p = 0.72, t-test, 2 sided; t Value: -0.36

6. Secondary Outcome: Change in Intent to Engage
Description: Intent to engage in health promotion was measured with an established scale (Ajzen, 1991) adapted for this project. The Intent To Engage questionnaire consists of eight questions each assessing assess intent, confidence and social support to complete health promotion activities. Each of these is rated on a likert-type scale ranging from 1-7 with some responses reverse scored so that higher responses indicate better intent, confidence, and social support. These are summed for a total score. Total scores range from 24 to 56.
Time Frame: Baseline and Follow-up
Population: Participants who completed both baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | -1.80 (12.99) | 3.10 (16.17)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = 0.88, t-test, 2 sided; t Value: 0.15

7. Secondary Outcome: Acceptability
Description: Measure of Patient self-report of acceptability of intervention. Participants responded to four questions using a 7 (0-7) point likert-type scale with higher ratings indicating higher acceptability. These were summed for a total score ranging from 0-28.
Time Frame: follow-up
Population: participants who completed follow-up measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | 23.9 (3.72) | 20.2 (5.20)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .08, t-test, 2 sided; t Value: 1.83

8. Secondary Outcome: New Health Behaviors From the Beginning of Classes Through Three Months Post End of Class
Description: A chart review was completed in order to identify documentation of new health behaviors. Mental health notes were first reviewed and then key terms were searched in all notes during the time period. S We considered a new health behaviors as: Starting or increasing physical activity in a formal program; Starting or increasing physical activity on own; Starting nicotine replacement/report cutting down or quitting smoking/join a smoking cessation group; Treatment for alcohol or SA/Report cutting down on Alcohol use; Report changing diet/formal nutrition consult/etc. Chart abstractors were instructed to make free text notes explaining each event the counted. These were reviewed by the PI for accuracy.
Time Frame: Start of class through 3 months post-class
Population: Veterans who completed both baseline and follow-up measures.
Measure: Number; unit: Events
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
Events | 17 | 7
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .16, Chi-squared — Chi Squared 1.98

9. Secondary Outcome: Change in CHAMPS (Community Healthy Activities Model Program for Seniors) Questionnaire for Older Adults - Physical Activity Duration
Description: Physical activity and cognitive/social activity will be measured by the CHAMPS (Stewart, et al., 2001) which asks respondents to identify if they participated in an activity (yes or no) how many times a week they participated (continuous variable) and if they did participate, for how many hours per week (rated on a 1 - 6 point scale ranging from less than one hour to more than 9 hours). The CHAMPS assesses for both physical and social/cognitive activities (e.g., "Visit with friends or family (other than those you live with);" "walk briskly").
Time Frame: baseline and 12 week follow-up
Population: participants who completed both baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | 1.85 (2.79) | 1.37 (4.06)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .85, t-test, 2 sided — t value: .19

10. Secondary Outcome: Change in CHAMPS (Community Healthy Activities Model Program for Seniors) Questionnaire for Older Adults - Cognitive Activity Frequency
Description: Physical activity and cognitive/social activity will be measured by the CHAMPS (Stewart, et al., 2001) which asks respondents to identify if they participated in an activity (yes or no) how many times a week they participated (continuous variable) and if they did participate, for how many hours per week (rated on a 1-6 point scale ranging from less than one hour to more than 9 hours). The CHAMPS assesses for both physical and social/cognitive activities (e.g., "Visit with friends or family (other than those you live with);" "walk briskly").
Time Frame: baseline and 12 week follow-up
Population: Participants who completed baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: times/week
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
times/week | -0.7 (5.48) | -2.0 (5.33)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .60, t-test, 2 sided — t value: .54

11. Secondary Outcome: Change in CHAMPS (Community Healthy Activities Model Program for Seniors) Questionnaire for Older Adults - Cognitive Duration
Description: as for outcome 10
Time Frame: baseline and 12 week follow-up
Population: Participants who completed baseline and follow-up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
units on a scale | -0.15 (3.72) | 1.99 (4.12)
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .26, t-test, 2 sided — t value: -1.17

12. Secondary Outcome: Number of Participants Beginning New Health Behaviors From the Beginning of Classes Through Three Months Post End of Class
Description: as for outcome 8
Time Frame: Start of class through 3 months post-class
Population: Veterans who completed both baseline and follow-up measures.
Measure: Number; unit: participants
Arm/Group | Get Moving and Get Well | Health and Humor Class
Number analyzed (Participants) | 10 | 10
participants | 8 | 5
Statistical Analysis 1: Comparison: Get Moving and Get Well vs Health and Humor Class; Test type: Superiority; p = .08, t-test, 2 sided — t value: 1.85

ADVERSE EVENTS:
Arm/Group | Get Moving and Get Well | Health and Humor Class
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/14
Other Adverse Events (participants affected / at risk) | 2/13 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Get Moving and Get Well (N=13) | Health and Humor Class (N=14)
Participant reproted Suicidal Ideation without Initent or Plan (Psychiatric disorders) | 0 (0) | 1 (1) — Veteran reported suicidal ideation. Licensed provider helped him return to emotional equilibrium. Veteran's primary mental health provider and bipolar support group leader were alerted. Veteran did attend the next classes with no problems reported.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Get Moving and Get Well (N=13) | Health and Humor Class (N=14)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Report of pain possibly related to class.
Displeasure with group (Psychiatric disorders) | 0 (0) | 1 (1) — Veteran became unhappy with compensation for time.

LIMITATIONS AND CAVEATS:
Due to small sample size, comparisons were completed descriptively to attempt to identify the emergence of trends. T-tests were used to assess for significant differences between groups and no significant differences were found.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes